CLINICAL TRIAL: NCT04859933
Title: AV Node Isolation in Atrial Fibrillation vs. Modulation by "Pace and Ablate" Strategy
Status: Completed | Type: Observational
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Sponsor
Other Study IDs: HDZ_ER_003_GI
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Atrial Fibrillation; AV Node Ablation; Escape; Rhythm
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AVNA group: Group of historical controls beeing treated with AV-node ablation
  Interventions: Procedure: AV-node ablation
- AVNI group: Inculudes all patients beeing treated with AV-node isolation
  Interventions: Procedure: AV-node isolation

INTERVENTIONS:
Procedure: AV-node isolation — Abaltion performed in the right atrium isolating the AV-node from the atrium
  Other Names: AVNI
  Groups: AVNI group
Procedure: AV-node ablation — Right sided ablation of the AV-node
  Other Names: AVNA
  Groups: AVNA group

SUMMARY:
AV-node ablation (AVNA) is a common therapy option for rate control strategy of permanent atrial fibrillation with numerous side effects. The investigators hypothesised that an isolation of the AV node is concomitant with less occurrence of new bundle brunch blocks, more frequent preservation and higher rate of escape rhythm compared to AVNA. This retrospective study includes 20 patients being treated with AV-node isolation (AVNI) and 40 historical AVNA-controls. Among others these two methods were compared regarding escape rhythm, delta QRS, procedure time, ablation points, fluoroscopy time and total dose area product (DAP).

ELIGIBILITY:
Inclusion Criteria:

* paroxysmal, persistend or permanent atrial fibrillation; indication for AVNA

Exclusion Criteria:

* other indications for AVNA than atrial fibrillation as AVNRT, atrial flutter, atrial tachycardia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Heart- and Diabetes Centre NRW for AV-node ablation/isolation.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
AV-node escape rhythm | intraoperative, follow-up after 1 to 3 month
bundle branch blocks | intraoperative, follow-up after 1 to 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Herz- und Diabeteszentrum NRW, Ruhr-Universität Bochum, Bad Oeynhausen, Germany

IPD SHARING:
Plan to Share IPD: No